CLINICAL TRIAL: NCT00115219
Title: A Multi-center, Randomized, Double-Blind, Active-Controlled Study Evaluating Efficacy and Safety of Etanercept 50 mg Twice Weekly (BIW) in Rheumatoid Arthritis Subjects Who Are Sub-optimal Responders to Etanercept 50 mg Once Weekly (QW)
Brief Title: Evaluating Efficacy and Safety of Etanercept 50 mg Twice Weekly (BIW) in Rheumatoid Arthritis (RA) Subjects Who Are Sub-Optimal Responders to Etanercept 50 mg Once Weekly (QW)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 20040275
Record Dates: First submitted 2005-06-21; First posted 2005-06-22 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-05

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis, RA; Enbrel® (etanercept); Clinical Trials, Amgen; Immunex, Methotrexate (MTX); Rheumatoid Arthritis (RA)
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept

INTERVENTIONS:
Drug: Etanercept

SUMMARY:
The purpose of this study objective will be to evaluate the efficacy and safety of etanercept 50 mg BIW in RA subjects who showed a sub-optimal response to standard dose etanercept (50 mg QW) and concomitant methotrexate therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Rheumatoid Arthritis
* RA with a disease duration > 6 months
* Current and prior but continuous etanercept (50 mg weekly) treatment for at least 5 months prior to screening
* Subjects must be receiving methotrexate (MTX) at a stable dose > 15 mg/week at least 4 weeks prior to screening
* Sub-optimal response to etanercept defined by the presence of the following criteria (based on 28 joint count) at screening: 5 or more swollen joints and 5 or more tender joints
* Subjects who are currently receiving oral corticosteroids must be on a dose equivalent to prednisone less than or equal to 10 mg/day at screening
* Subjects who are currently receiving non-steroidal anti-inflammatory drugs (NSAIDs), must be on a stable dose for at least 2 weeks prior to screening
* Subjects who are currently receiving DMARD therapy (including sulfasalazine, hydroxy-chloroquine and leflunomide), must be on a stable dose for at least 4 weeks prior to screening

Exclusion Criteria:

* Nursing mothers, female subjects planning on becoming pregnant, or male subjects planning a pregnancy with their spouse/partner while in the study
* ACR functional class IV
* Receipt of any investigational drug or biologic within 4 weeks of study drug initiation
* Concurrent or history of psychiatric disease that would interfere with ability to comply with study protocol or give informed consent
* History of alcohol or drug abuse within 12 months of screening visit
* Severe comorbidities including: History of cancer (other than resected cutaneous basal and squamous cell carcinoma, and in situ cervical cancer) within 5 years of screening visit. Documentation of disease-free state since treatment required; Diagnosis of Class III or IV congestive heart failure (CHF) or myocardial infarction (MI) within 12 months of screening; Unstable or stable angina pectoris; Uncontrolled hypertension (defined as systolic blood pressure measurement of greater than 180 mm Hg or a diastolic blood pressure of greater than 110 mm Hg); Oxygen-dependent pulmonary disease; Known HIV-positive status or other immunodeficiency syndromes; Chronic hepatitis B (HbsAg) or C (HCV); Systemic lupus erythematosus (SLE); CNS demyelinating events suggestive of multiple sclerosis; Presence of active infection or any underlying diseases that could predispose subjects to infection (e.g., history of recurrent infections, non-healing leg ulcers, advanced or poorly controlled diabetes); Active or prior history of tuberculosis (or known exposure).
* Concurrent treatment with cyclophosphamide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2005-05

PRIMARY OUTCOMES:
Proportion of subjects achieving a good or moderate DAS28 response (as defined by the EULAR28 response criteria) at Week 12

SECONDARY OUTCOMES:
Proportion of subjects who achieve American College of Rheumatology (ACR) 20, 50, and 70 responses at Weeks 12 and 24
Proportion of subjects achieving a good or moderate DAS28 response (as defined by the EULAR28 response criteria at Week 24 and the proportion achieving clinical remission (DAS28<2.6) at Weeks 12 and 24
Changes from baseline with respect to the DAS28 score and ACR score (including HAQ) criteria at Weeks 12 and 24
Changes from baseline in patient-reported outcomes as measured by the SF-36 at Weeks 12 and 24
Proportion of etanercept 50mg BIW responders at Week 12 who mantain a clinical improvement with etanercept 50mg QW (defined as no DAS28 increase of greater than 0.6 from Week 12) at Week 24
Safety (SAEs and AEs) in three study periods (4-week open label run-in period, 12-week double blinded period A, and 12-week open-label period B)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Weinblatt ME, Schiff MH, Ruderman EM, Bingham CO 3rd, Li J, Louie J, Furst DE. Efficacy and safety of etanercept 50 mg twice a week in patients with rheumatoid arthritis who had a suboptimal response to etanercept 50 mg once a week: results of a multicenter, randomized, double-blind, active drug-controlled study. Arthritis Rheum. 2008 Jul;58(7):1921-30. doi: 10.1002/art.23493. PMID 18576334
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_916_ENBREL_20040275.pdf
- See also: FDA-approved Drug Labeling — http://www.enbrel.com
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com